CLINICAL TRIAL: NCT04964622
Title: Effect of Preoperative Single Dose of Sodium Ibuprofen Versus Placebo on Post-operative Pain for Patient With Symptomatic Irreversible Pulpitis Related to Mandibular Molar Teeth: Double Blind Randomized Controlled Trial
Brief Title: the Effect of Preoperative Sodium Ibuprofen on Postoperative Endodontic Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samah Sobhie Abdalla, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: postoperative endodontic pain
Record Dates: First submitted 2021-07-01; First posted 2021-07-16 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Irreversible Pulpitis
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: patient with symptomatic irriversible pulpitis
Who Masked: Participant, Care Provider
Masking Description: drug will be put in sealed envelop and assistant supervisor will generate random sequence
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nurofen (Other): sodium ibuprofen 1 tablet (256) 30 minutes before treatment administered once (oral)
  Interventions: Drug: nurofen
- placebo (Placebo Comparator): starch tablet 30 minutes before treatment administered once (oral)
  Interventions: Drug: nurofen

INTERVENTIONS:
Drug: nurofen — tablet
  Other Names: sodium ibuprofen

SUMMARY:
The aim of this study is to clinically compare post-operative pain levels after administration of preoperative single dose of sodium ibuprofen versus placebo for patient with symptomatic irreversible pulpitis related to mandibular molar teeth.

DETAILED DESCRIPTION:
Oral pharmacologic agents have been the primary option, and the use of drugs has increased exponentially. Many pharmacological agents have been used to manage endodontic pain, including Non-steroidal Anti-inflammatory Drugs (NSAIDs),.administration of NSAIDs before root canal treatment will reduce inflammatory process before it begins. NSAIDs are widely used to control post endodontic pain They act by blocking the activity of cyclooxygenase (COX 1 and 2) enzyme. In human dental pulps with irreversible pulpitis, a higher level of expression of COX 2.In cases of irreversible pulpitis NSAIDS can be administered preoperatively since they reduce the level of prostaglandinE2(PGE2) which is responsible for sensitization of nociceptors. Ibuprofen is one of the most commonly used NSAIDs and a potent inhibitor of prostaglandin (PG) synthesis that can manage various pain types and has anti-inflammatory activity. Enhancements in ibuprofen acid's pharmacokinetics have led to the development of ibuprofen salts with a faster dissolution rate and onset of action. These ibuprofen salts.Fast acting ibuprofen like Sodium ibuprofen delivers maximum plasma drug concentrations at about 30-40 min, compared with around 90-120 min for standard ibuprofen acid formulations

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years old and below 66.
* Male or female
* Patients seeking root canal treatment
* Mandibular posterior molarteeth with Symptomatic irreversible pulpitis .
* Spontaneous pain
* Systematically healthy patient(ASA I,II)

Exclusion Criteria:

* Medically compromised patients having significant systemic disorders. (ASA III or IV)
* History of intolerance to NSAIDS.
* Patients with two or more adjacent teeth requiring endodontic treatment.
* External root resorption
* Internal root resorption
* Vertical root fracture
* Periapical lesion
* Pregnancy
* Use of ibuprofen in the last 12 hour
* Bleeding disorder
* Long term corticosteroid use
* Mobility Grade II or III.
* Pocket depth more than 5mm.
* Previous root canal therapy.
* Non-restorability
* Temporomandibular joint (TMJ) problems, bruxism, clenching or traumatic occlusion.
* Inability to perceive the given instructions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | Post-operative pain will be assessed immediately after treatment ,at 6 hours, at 12 hours, at 24 hours and 48 hours
  pain will be measured by visual analogue scale(VAS). Postoperative pain levels were documented by the patients immediately after obturation, 6, 12, 24 and 48 hours post-treatment. The VAS consists a 10-cm line anchored by 2 extremes, ''no pain'' and ''pain as bad as it could be.'' Patients were asked to make a mark on the line that represents their level of perceived pain. Readings were transformed into categories; no pain (range of 0-4mm), mild pain (range of 5-44mm), moderate pain (range of 45-74mm) and severe pain (range of 75-100mm)

SECONDARY OUTCOMES:
need for rescue medication | Amount of analgesics taken by the patient after root canal treatment, up to 48 hours postoperatively
  Amount of analgesics taken by the patient after root canal treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Smith EA, Marshall JG, Selph SS, Barker DR, Sedgley CM. Nonsteroidal Anti-inflammatory Drugs for Managing Postoperative Endodontic Pain in Patients Who Present with Preoperative Pain: A Systematic Review and Meta-analysis. J Endod. 2017 Jan;43(1):7-15. doi: 10.1016/j.joen.2016.09.010. Epub 2016 Dec 6. PMID 27939729
- [Result] Suresh N, Nagendrababu V, Koteeswaran V, Haritha JS, Swetha SD, Varghese A, Natanasabapathy V. Effect of preoperative oral administration of steroids in comparison to an anti-inflammatory drug on postoperative pain following single-visit root canal treatment - a double-blind, randomized clinical trial. Int Endod J. 2021 Feb;54(2):198-209. doi: 10.1111/iej.13416. Epub 2020 Nov 12. PMID 32976660